CLINICAL TRIAL: NCT06176586
Title: Investigating the Effects of Mat Pilates Exercises in Patients With Axial Psoriatic Arthritis
Brief Title: Mat Pilates Exercise Program in Patients With Axial Psoriatic Arthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Deniz Bayraktar, Assistant Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSApilex
Record Dates: First submitted 2023-12-07; First posted 2023-12-19 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Psoriatic Arthritis
Keywords: Pilates Exercise; Arthritis; Spine Mobility
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Progressive mat Pilates exercises will be administered to by a physiotherapist in addition to the routine medical treatment.
  Interventions: Other: Mat Pilates Exercises
- Control Group (No Intervention): Patients in control group will not receive any exercise intervention. They will continue to their routine medical treatment.

INTERVENTIONS:
Other: Mat Pilates Exercises — The intervention will consist of mat Pilates exercises performed twice a week over a duration of 12 weeks, as an adjunct to the routine medical treatment for the patients, under the guidance of a qualified physiotherapist. Each exercise session will last for approximately 60 minutes. The treatment protocol will encompass targeted mobility exercises for the thoracic and lumbar regions, along with strengthening exercises focusing on core activation. The exercise program will be progressed in every four weeks.
  Arms: Exercise Group

SUMMARY:
The aim of this study is to investigate the effectiveness of mat Pilates exercises on spinal mobility, spinal muscle endurance, disease activity, fatigue, emotional well-being, physical performance, and overall quality of life in Psoriatic Arthritis (PsA) patients with axial involvement.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease commonly accompanied by joint involvement known as psoriatic arthritis (PsA) [1]. PsA is a subgroup of spondyloarthritis and is characterized by peripheral arthritis, dactylitis, enthesitis and spondylitis. Axial involvement, which occurs in approximately 40% of PsA patients may affect the entire spine, particularly the sacroiliac joint, leading to reduced cervical rotation, lateral flexion and anterior flexion of the spine [2,3]. Exercise interventions in PsA primarily aim to relieve pain, improve mobility and enhance functional capacity [4]. Mat Pilates exercises have been demonstrated as a safe and beneficial intervention in various rheumatic diseases, exhibiting significant improvements in functional status, fatigue, disease activity, pain, and overall quality of life [5-7]. Additionally, Pilates has been reported as effective in maintaining and enhancing spinal mobility [8,9]. However, despite these favorable outcomes, the efficacy of Pilates exercises in PsA remains unexplored.

The aim of this study is to investigate the effectiveness of mat pilates exercises in psoriatic arthritis patients with axial involvement.

ELIGIBILITY:
Inclusion Criteria:

* Being classified as PsA according to CASPAR Classification Criteria
* Being between the ages of 18-65
* Volunteering to participate in the study

Exclusion Criteria:

* Any additional systemic disease other than PsA
* Any other condition that may prevent participation/continuation of the exercise program or completion of the assessments
* Regular exercise habits (following a structured exercise program at least 3 days a week)
* Being included in a physiotherapy and rehabilitation program within the last 6 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Performance | At baseline and 12 weeks later
  The Ankylosing Spondylitis Performance Index (ASPI) will be used. The ASPI consists of three physical performance tasks: (a) bending forward to pick up six pencils from the floor; (b) putting on socks (average of three repetitions); and (c) getting up from the floor (average of three repetitions). Time to complete a task will be recorded in seconds for each test.

SECONDARY OUTCOMES:
Change in Functional Status | At baseline and 12 weeks later
  Bath Ankylosing Spondylitis Functional Index (BASFI) will be used. This self-reported scale evaluates the degree of functional limitation of patients in activities of daily living. It consists of 10 questions scored between 0-10 (0: easy, 10: impossible). The higher total scores indicate more functional limitation.
Change in Trunk Muscle Endurance | At baseline and 12 weeks later
  A static endurance test (lateral bridge test) will be employed to evaluate trunk muscle endurance. During this assessment, patients will be positioned in side-lying. Participants will be required to maintain this lateral bridge position for as long as possible, and the duration until the position cannot be maintained will be recorded in seconds.
Change in Spinal Mobility | At baseline and 12 weeks later
  Spinal mobility will be assessed by using the Bath Ankylosing Spondylitis Mobility Index including cervical rotation, modified Schober test (anterior flexion of the spine), maximal intermalleolar distance, lateral flexion of the spine, and tragus-wall distance. Higher scores indicate more limited spinal mobility.
Chance in Disease Activity | At baseline and 12 weeks later
  The Disease Activity Index for Psoriatic Arthritis (DAPSA) will be used for evaluating the disease activity. DAPSA is a composite score including the number of tender joints (over 68 joints), the number of swollen joints (over 68 joints), C-Reactive protein (CRP) level, the patient's self-reported health status, and evaluation of the patient's health status by the physician. DAPSA is calculated by summing all the values, and higher scores indicate higher disease activity.
Change in Fatigue | At baseline and 12 weeks later
  The Fatigue Severity Scale (FSS) will be used to evaluate the fatigue. It comprises 9 items that assess the severity of fatigue symptoms experienced by participants over the previous week. Each question is scored on a scale ranging from 1 (strongly disagree) to 7 (strongly agree), and the scores are then averaged to derive the total score. Higher scores indicate more fatigue.
Change in Emotional Status | At baseline and 12 weeks later
  The Hospital Anxiety and Depression Scale (HADS) will be used to evaluate emotional status. The HADS includes two sections: depression (7 questions) and anxiety (7 questions). Each question is scored between 0 and 3. Higher scores indicate higher anxiety or depression levels.
Change in Quality of Life | At baseline and 12 weeks later
  The Psoriatic Arthritis Quality of Life (PsAQoL) questionnaire will be used to assess the disease-related changes in quality of life. The PsAQoL includes 20 questions, each answered with either yes (1 point) or no (0 point). Higher scores indicate a reduced quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Bayraktar, PhD, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data may only be provided upon a reasonable request for academic research purposes.

REFERENCES:
- [Background] Parisi R, Symmons DP, Griffiths CE, Ashcroft DM; Identification and Management of Psoriasis and Associated ComorbidiTy (IMPACT) project team. Global epidemiology of psoriasis: a systematic review of incidence and prevalence. J Invest Dermatol. 2013 Feb;133(2):377-85. doi: 10.1038/jid.2012.339. Epub 2012 Sep 27. PMID 23014338
- [Background] Ogdie A, Weiss P. The Epidemiology of Psoriatic Arthritis. Rheum Dis Clin North Am. 2015 Nov;41(4):545-68. doi: 10.1016/j.rdc.2015.07.001. Epub 2015 Sep 11. PMID 26476218
- [Background] Gladman DD, Antoni C, Mease P, Clegg DO, Nash P. Psoriatic arthritis: epidemiology, clinical features, course, and outcome. Ann Rheum Dis. 2005 Mar;64 Suppl 2(Suppl 2):ii14-7. doi: 10.1136/ard.2004.032482. PMID 15708927
- [Background] Chimenti MS, Triggianese P, Conigliaro P, Santoro M, Lucchetti R, Perricone R. Self-reported adherence to a home-based exercise program among patients affected by psoriatic arthritis with minimal disease activity. Drug Dev Res. 2014 Nov;75 Suppl 1:S57-9. doi: 10.1002/ddr.21197. PMID 25381979
- [Background] Altan L, Korkmaz N, Dizdar M, Yurtkuran M. Effect of Pilates training on people with ankylosing spondylitis. Rheumatol Int. 2012 Jul;32(7):2093-9. doi: 10.1007/s00296-011-1932-9. Epub 2011 Apr 17. PMID 21499876
- [Background] Caglayan BC, Keskin A, Gur Kabul E, Basakci Calik B, Bas Aslan U, Karasu U. Effects of clinical Pilates exercises in individuals with fibromyalgia: A randomized controlled trial. Eur J Rheumatol. 2021 Jul;8(3):150-155. doi: 10.5152/eurjrheum.2020.20037. PMID 33372888
- [Background] Acar Y, Ilcin N, Gurpinar B, Can G. The effects of clinical pilates training on disease-specific indices, core stability, and balance in patients with ankylosing spondylitis. J Bodyw Mov Ther. 2023 Jan;33:69-75. doi: 10.1016/j.jbmt.2022.09.010. Epub 2022 Sep 23. PMID 36775528
- [Background] Oksuz S, Unal E. Comparison of the effects of aerobic training alone versus aerobic training combined with clinical Pilates exercises on the functional and psychosocial status of patients with ankylosing spondylitis: A randomized controlled trial. Physiother Theory Pract. 2023 Jan;39(1):61-71. doi: 10.1080/09593985.2021.2005199. Epub 2021 Nov 18. PMID 34791973